CLINICAL TRIAL: NCT02117427
Title: Safety and Efficacy of Sustained Erythropoietin Therapy of Anemia in Chronic Kidney Disease (CKD) Patients and End-Stage Renal Disease (ESRD) Dialysis Patients Using MDGN201 TARGTEPO
Brief Title: TARGTEPO Treatment for Anemia in Chronic Kidney Disease (CKD) Patients and End-Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Collaborators: Medgenics Medical Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MG-EP-RF-02
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-02

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): MDGN201 TARGTEPO secreting EPO (18-25 IU/Kg/day)
  Interventions: Biological: MDGN201 TARGTEPO
- Group B (Experimental): MDGN201 TARGTEPO secreting EPO (35-45 IU/Kg/day)
  Interventions: Biological: MDGN201 TARGTEPO
- Group C (Experimental): MDGN201 TARGTEPO secreting EPO (55-65 IU/Kg/day)
  Interventions: Biological: MDGN201 TARGTEPO

INTERVENTIONS:
Biological: MDGN201 TARGTEPO — Erythropoietin secreted by TARGTEPO transduced with MDGN201

SUMMARY:
The objectives of this study are to assess safety and to evaluate the biologic activity of TARGTEPO treatment.

DETAILED DESCRIPTION:
This is a Phase I-II, open-label study. Each patient will receive targeted dose of EPO delivered via TARGTEPO. The targeted doses will be determined according to 3 cohorts as follows: Group A (18-25 IU/Kg/day), Group B (35-45 IU/Kg/day), Group C (55-65 IU/Kg/day). The objective is to evaluate safety and biologic activity of TARGTEPO treatment when maintaining Hb levels within the target range of 9-12 g/dl. Biological activity assessments will include duration of TARGTEPO secretion as measured by serum EPO levels above baseline

ELIGIBILITY:
Inclusion Criteria:

1. For ESRD patients: Subject diagnosed with Anemia due to Chronic Renal Failure CKD stage 5 on hemodialysis treatment for at least 6 months. Average Hb during last month between 9 to 12g/dL.
2. Kt/V >1
3. INR not higher than 1.2
4. Serum albumin >3.5
5. Subjects with adequate iron stores (transferrin saturation > 20.0% and/or ferritin >100 ng/ml).

Exclusion Criteria:

1. Uncontrolled hypertension (defined as diastolic blood pressure > 110 mmHg or systolic blood pressure > 180 mmHg during screening).
2. Subjects who receive oral anti-coagulation treatment (e.g. warfarin)
3. Subjects who receive Acetyl Salicylic Acid (ASA) above 325 mg/day or patients who receive ASA treatment between 100mg/d and 325 mg/d who cannot discontinue it for 1 week prior to each EPODURE procedure
4. Patients currently receiving injections of long-acting Erythropoiesis Stimulating Agents (ESA) (e.g. Aranesp, Mircera), a patient on long acting ESA can be switched to a short acting preparation (e.g Eprex) and enroll in the study after meeting the inclusion criteria and not meeting any other exclusion criteria.
5. Congestive heart failure (New York Heart Association functional class III or IV).
6. Grand mal seizures within 2 years of the screening visit.
7. Clinical evidence of severe hyperparathyroidism as defined by PTH levels of > 10 times the upper normal limits.
8. Major surgery within 12 weeks of the screening visit.
9. Systemic hematologic diseases (e.g., sickle cell anemia, thalassemia, myelodysplastic syndromes, hematologic malignancy, myeloma, hemolytic anemia).
10. Current systemic infection, active inflammatory disease, or malignancy under active treatment.
11. Subjects known to have tested positive at any time in the past for antibodies to erythropoietic proteins.
12. Subject has history of malignancy within the past 2 years prior to the screening visit, with the exception of basal cell carcinoma.
13. Subjects with other concurrent severe and/or uncontrolled medical condition which could compromise participation in the study (i.e. active infection, uncontrolled diabetes, uncontrolled hypertension, congestive heart failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, uncompensated cirrhosis, active upper GI tract ulceration).
14. Subject is currently enrolled in, or has not yet completed a period of at least 30 days or five half-lives of the investigational drug whichever is longer, since ending other investigational device or drug trial(s) prior to Screening phase.
15. Psychiatric, addictive, or any other disorder that compromises ability to provide informed consent for participation in this study.
16. Female subjects of child-bearing potential and males that do not agree to use acceptable methods of contraception during the study.
17. Pregnant and lactating female subjects.
18. Chronic alcoholic or drug abuse subjects.
19. Steroid or other immunosuppressive treatment (other than topical or inhaled steroids).
20. Subjects unwilling or unable to comply with the study procedures.
21. EPO Naïve subjects.
22. Known sensitivity to Gentamycin and Amphotericin
23. History of chronic or active Hepatitis B and/or C infection or positive serology at screening and known positive HIV or positive serology at screening.
24. Subject had blood transfusion within 84 days prior to Screening visit.
25. Subject has a date for renal transplantation.
26. Subject has a temporary or permanent hemodialysis catheter, unless: Subject has a permanent hemodialysis catheter over 6 months without signs/events of line sepsis.
27. Refer to the USPI - Depo-Medrol - Methylprednisolone Acetate - Injectable (Appendix A) for any concomitant drug taken by the patient which its interaction with Depo-Medrol will warrant exclusion from this protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shany Blum, MD PhD, Study Director — Aevi Genomic Medicine, LLC, a Cerecor company
Locations (5):
- Israel (5):
  - Barzili Medical Center, Ashkelon
  - Meir Medical Center, Kfar Saba
  - Medical Center of the Galilee, Nahariya
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Zrifin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.nejm.org/doi/full/10.1056/NEJMc1606202

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 14 patients signed the Informed Consent Form and underwent the study screening procedures. Of these 14 patients, a total of 11 patients were enrolled into Study MG-EP-RF-02. These 11 patients are included in the ITT cohort. One patient (Group B) had an SAE prior to study procedures and became no longer eligible.
Period: Overall Study
Arm/Group | Group A: 18-25 IU/Kg/Day | Group B: 35-45 IU/Kg/Day | Group C: 55-65 IU/Kg/Day
Started | 6 | 5 | 0
Run in Phase & Harvest | 6 | 4 | 0
Implantation & Efficacy | 6 | 4 | 0
Safety Follow-up | 1 | 0 | 0
Long Term Safety Follow-up | 1 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 5 | 5 | 0
Not completed — Permanent need for exogenous EPO Tx | 2 | 0 | 0
Not completed — Permanent need for exogenous ESA Tx | 3 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0
Not completed — No longer meets inclusion criteria | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: 18-25 IU/Kg/day
- Group B: 35-45 IU/Kg/day
- Group C: 55-65 IU/Kg/day
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 6 | 5 | 0 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 0 | 6
  >=65 years | 4 | 1 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 4 | 4 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 5 | 4 | 0 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total EPO Secretion
Time Frame: up to 52 weeks
Population: Due to the small sample size and the dispersion of total EPO secretion, the efficacy analyses were performed on all of the patients as a single cohort of intended dose between 25 and 45 U/Kg/d. One subject enrolled was discontinued prior to study procedures and became no longer eligible.
Measure: Mean (Full Range); unit: U/Kg/d
Arm/Group | All Subjects Enrolled
Number analyzed (Participants) | 10
U/Kg/d | 24.1 [16.5 to 50.8]

2. Primary Outcome: Percent (%) of Hb Measurements After Implantation Within 9-11 g/dL
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: percent
Arm/Group | All Subjects Enrolled
Number analyzed (Participants) | 10
percent | 49.2 [1.7 to 88.1]

3. Primary Outcome: Percent (%) of Hb Measurements After Implantation Within 9-12 g/dL
Description: Due to the small sample size and the dispersion of total EPO secretion, the efficacy analyses were performed on all of the patients as a single cohort of intended dose between 25 and 45 U/Kg/d.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: percent
Arm/Group | All Subjects Enrolled
Number analyzed (Participants) | 10
percent | 75.3 [25.0 to 88.1]

ADVERSE EVENTS:
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/6 | 4/4 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=6) | Group B (N=4) | Group C (N=0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=6) | Group B (N=4) | Group C (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoparathyroidism secondary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal microaneurysm NOS (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (11) | 3 (8) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (15) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysthymic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (5) | 1 (4) | 0 (0)
Hypotension (Vascular disorders) | 3 (12) | 1 (3) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should the investigator wish to publish the results of this study, the investigator agrees to provide Medgenics with a manuscript for review 60 days prior to submission for publication. Medgenics retains the right to delete from the manuscript information that is confidential and proprietary and to object to suggested publication and/or its timing (at the Company's sole discretion).